CLINICAL TRIAL: NCT05937516
Title: Guidewire Use for Nasopharyngeal Passage in Pediatric Nasotracheal Intubation: A Randomized Prospective Study
Brief Title: Guidewire Use in Nasotracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Asım Esen, Assistant Professor ASIM ESEN, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: a.esen001
Record Dates: First submitted 2023-06-20; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Epistaxis Nosebleed; Pharyngeal Bleeding
Keywords: Airway management; Intubation complication; Nasotracheal intubation; Nasal bleeding
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: After intubation was completed, bleeding was evaluated by the other investigator who did not know the patient's group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Sham Comparator): Nasotracheal intubation will be applied conventionally to patients in this group.
  Interventions: Device: Nasotracheal intubation with conventionally
- Study Group (Active Comparator): In the study group (Group S), a guide wire will be inserted into the ETT before intubation and angled 100-120 degrees to the distal end (in the shape of a hockey stick). The angulation will not be sharp but slightly curved and the apex of the angulation will be 2.5-3 cm proximal from the distal end. The ETT will be positioned perpendicular to the face and inserted into the nostril. After the angled part of the ETT passes through the nostrils, it will be directed to caudally according to the angle given to the tip of the ETT. Meanwhile, the ETT will be moved as a whole to prevent the ETT tip from contacting the posterior wall of the nasopharynx. When the ETT tip reaches the oropharynx, the guidewire will be removed and the rest of the intubation will be completed as in the conventional method.
  Interventions: Device: Nasotracheal intubation with angled ETT using guidewire

INTERVENTIONS:
Device: Nasotracheal intubation with conventionally — Nasotracheal intubation will be applied conventionally to patients in this group.
  Arms: Control Group
Device: Nasotracheal intubation with angled ETT using guidewire — a guide wire will be inserted into the ETT before intubation and angled 100-120 degrees to the distal end (in the shape of a hockey stick). The angulation will not be sharp but slightly curved and the apex of the angulation will be 2.5-3 cm proximal from the distal end. The ETT will be positioned perpendicular to the face and inserted into the nostril. After the angled part of the ETT passes through the nostrils, it will be directed to caudally according to the angle given to the tip of the ETT. Meanwhile, the ETT will be moved as a whole to prevent the ETT tip from contacting the posterior wall of the nasopharynx. When the ETT tip reaches the oropharynx, the guidewire will be removed and the rest of the intubation will be completed as in the conventional method.
  Arms: Study Group

SUMMARY:
During nasotracheal intubation, nasopharyngeal trauma and associated bleeding may occur. The investigators think that some of this bleeding is due to trauma to the posterior wall of the nasopharynx. The investigators designed this study, thinking that if nasopharyngeal posterior wall trauma can be prevented, some of these bleedings can be prevented.

DETAILED DESCRIPTION:
Nasotracheal intubation (NTI) is a frequently used airway management method in pedodontic dental treatments performed under general anesthesia. However, nasopharyngeal trauma and associated bleeding are common during conventional NTI. In this study, the investigators aimed to examine the effect of angling the end of the endotracheal tube (ETT) by placing a guide wire inside the ETT on nasopharyngeal bleeding.

The patients included in the study were randomized into two groups. In the control group (Group C), NTI will be done conventionally. In the study group (Group S), a guide wire will be inserted into the ETT before intubation and angled 100-120 degrees to the distal end (in the shape of a hockey stick). The angulation will not be sharp but slightly curved and the apex of the angulation will be 2.5-3 cm proximal from the distal end. The ETT will be positioned perpendicular to the face and inserted into the nostril. After the angled part of the ETT passes through the nostrils, it will be directed to caudally according to the angle given to the tip of the ETT. Meanwhile, the ETT will be moved as a whole to prevent the ETT tip from contacting the posterior wall of the nasopharynx. When the ETT tip reaches the oropharynx, the guidewire will be removed and the rest of the intubation will be completed as in the conventional method.

ELIGIBILITY:
Inclusion Criteria:

* 2-12 years old
* American Society of Anesthesiologists I-III
* Patients with elective dental surgery
* Patients whose parents have accepted informed consent forms
* Patients without previous nasopharyngeal anomalies
* Patients without previous nasopharyngeal surgeries
* Patients without upper airway infections

Exclusion Criteria:

* Under 2 or over 12 years old
* Emergency surgeries
* Patients whose parents have not accepted informed consent forms
* Patients with previous nasopharyngeal anomalies
* Patients with previous nasopharyngeal surgeries
* Patients with upper airway infections

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Presence of blood in oropharynx or on the endotracheal tube | In the first minute after intubation
  The presence of blood in the oropharynx or endotracheal tube will be defined by assessing it on a scale. (0 = no blood, 2 = mild, that is, dye-like blood on the endotracheal tube, 3 = severe, that is, obvious blood in the oropharynx).
Presence of blood in oropharynx or on the endotracheal tube | In the fifth minute after intubation
  The presence of blood in the oropharynx or endotracheal tube will be defined by assessing it on a scale. (0 = no blood, 2 = mild, that is, dye-like blood on the endotracheal tube, 3 = severe, that is, obvious blood in the oropharynx).

CONTACTS AND LOCATIONS:
Overall Officials: asim esen, Asst Prof, Principal Investigator — Bezmialem Vakif University, Faculty of Medicine
Locations (1):
- Bezmialem Vakif University, Faculty of Medicine, Fatih, Istanbul, Turkey (Türkiye)